CLINICAL TRIAL: NCT02166593
Title: A Study to Evaluate the Efficacy and Safety of Pravastatin/Fenofibrate Complex in Patients With Combined Dyslipidemia With Adequately Controlled LDL-C But Inadequately Controlled Triglyceride Level by Atorvastatin Monotherapy
Brief Title: Clinical Trial to Evaluate the Efficacy and Safety of Pravafenix Cap to Verify the Superiority Than Atorvastatin
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Yooyoung Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: YYP-Pravafenix-C31301
Record Dates: First submitted 2014-05-27; First posted 2014-06-18 (Estimated); Last update posted 2018-09-28 (Actual); Status verified 2018-09

CONDITIONS: Combined Dyslipidemia
MeSH Terms: interventions — Atorvastatin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Pravastatin 40mg/Fenofibrate160mg (Experimental): Pravastatin (40mg/day) Fenofibrate (160mg/day)
  Interventions: Drug: Pravastatin40mg/Fenofibrate160mg; Drug: Atorvastatin Sodium 10mg
- Atorvastatin Sodium (Active Comparator): Atorvastatin Sodium (10mg/day)
  Interventions: Drug: Pravastatin40mg/Fenofibrate160mg; Drug: Atorvastatin Sodium 10mg

INTERVENTIONS:
Drug: Pravastatin40mg/Fenofibrate160mg — Pravafenix(Pravastatin40mg/Fenofibrate160mg)
  Other Names: Pravafenix(Pravastatin40mg/Fenofibrate160mg)
Drug: Atorvastatin Sodium 10mg — Lipitor 10mg(Atorvastatin Sodium)
  Other Names: Lipitor 10mg(Atorvastatin Sodium)

SUMMARY:
1. Target disease : Patients with combined dyslipidemia with adequately controlled LDL-C but inadequately controlled triglyceride level by atorvastatin monotherapy
2. Study objective : The objective of this study is to demonstrate that Pravafenix Cap. is clinically superior to atorvastatin by evaluating a percent change in Non-HDL-C in each group after 8 weeks treatment with atorvastatin or Pravafenix Cap. (pravastatin sodium/fenofibrate) in patients with adequately controlled LDL-C but inadequately controlled triglyceride level by atorvastatin monotherapy in a multicenter, randomized, double blind setting.
3. Phase and design : A multicenter, double blind, randomized, active controlled, parallel-design, Phase 3 study
4. Duration of study : 12 months from the IRB approval date
5. Duration of administration : 4-week single blind run-in period plus 8-week double blind treatment period

DETAILED DESCRIPTION:
This study is to Evaluate the Efficacy and Safety of Pravastatin/Fenofibrate Complex in Patients With Combined Dyslipidemia With Adequately Controlled LDL-C But Inadequately Controlled Triglyceride Level by Atorvastatin Monotherapy. After administrating the atorvastatin or Pravafenix Cap. (pravastatin sodium/fenofibrate) for 8 weeks, evaluate the variation of the Non-HDL-C for each arm. Ultimatly verificaite the Pravafenix Cap. (pravastatin sodium/fenofibrate) have better effects than atorvastatin.

ELIGIBILITY:
Inclusion Criteria:

Screening visit (Pre-Study Visit :D-28)

1. Men and women at the age ≥ 20 and < 80
2. Patients at a high risk of coronary heart disease according to the NCEP ATPIII guidelines

   * Patients with coronary artery disease, or
   * Patients with symptomatic carotid artery disease, or
   * Patients with peripheral vascular disease, or
   * Patients with abdominal aneurysm, or
   * Patients with diabetes mellitus, or
   * Patients at a more than 20% 10-year risk of coronary heart disease, or
3. LDL-C < 160mg/dL at screening
4. Fasting triglyceride (TG) level ≥ 150mg/dL and < 500mg/dL at screening
5. HDL-C level <40mg/dL (Male Patient), <50mg/dL(Female Patient)
6. Voluntary written informed consent to study participation

Secondary visit (Visit 2 (D0))

1. LDL-C < 100mg/dL after the 4-week atorvastatin run-in period
2. Fasting TG level ≥ 150mg/dL and < 500mg/dL after the 4-week atorvastatin run-in period
3. HDL-C level <40mg/dL (Male Patient), <50mg/dL(Female Patient)

Exclusion Criteria:

1. Acute arterial disease (history of unstable angina pectoris, myocardial infarction, acute coronary syndrome, transient ischemic attack, cerebrovascular disease, coronary bypass, or coronary artery disease within 3 months prior to study participation)
2. Revascularzation procedure or aortic aneurysm operation within 6 months prior to study participation
3. Myopathy, history of rhabdomyolysis or myopathy due to statins or fibrates, or elevated CK level ≥ 5 x upper limit of normal (ULN) during the previous statin treatment
4. Acute or chronic pancreatitis due to hypertriglyceridemia
5. Cardiovascular, hepatic, neurological, endocrine, or other serious systemic disease that may affect the study conduct or interpretations of the study results
6. Known positive serum tests to human immunodeficiency virus (HIV) Antibody I or II
7. Diagnosis of cancer within the past 2 years (except successfully treated basal cell carcinoma and squamous cell carcinoma)
8. Patients treated with prohibited concomitant medications during the study period or those for whom treatment with prohibited concomitant medications is considered inevitable (systemic or inhalant corticosteroids may be allowed during the study provided that the treatment is maintained at the same dose.)
9. Administration of or will be administered with periodic sex hormone therapies or oral contraceptives within 2 months prior to the screening visit or during the study participation
10. Moderate to severe renal impairment (GFR<60ml/min) at screening
11. Severe hepatic impairment with AST/ALT level > 3 x ULN at screening (biliary cirrhosis, active liver disease, or continued increases in transaminases by unknown causes (> 3 x ULN), etc.)
12. Uncontrolled hypothyroidism
13. Uncontrolled diabetes mellitus (HbA1c>8.5%)
14. Hyperlipidemia Class I, IIa, IV, or V
15. Requiring insulin treatment for diabetes mellitus
16. Allergies or hypersensitivity reactions to the study drug
17. Patients known to have, or suspected of having a history of drug or alcohol abuse within the past 2 years
18. Confirmed pregnant or lactating women at screening
19. Women of childbearing potential at screening and planning to become pregnant during the study. Women at the childbearing age who did not undergo surgical sterilization may participate in the study only if the pregnancy test is determined negative and should maintain effective contraceptive methods throughout the study period. Periodic abstinence (e.g., calendar method, ovulation method, symptothermal method, post-ovulation method) and self control are not considered to be acceptable contraceptive methods, and use of hormonal contraceptives is not allowed.
20. Having participated in another clinical trial within 1 month prior to screening
21. History of photoallergic or phototoxic reactions during treatment with fibrates or ketoprofen
22. Biliary disease
23. Interstitial pulmonary disease
24. Other patients considered by the principal investigator or sub-investigator inappropriate for study participation

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 302 (Actual)
Dates: Start 2014-05; Primary Completion 2018-01 (Actual); Study Completion 2018-01 (Actual)

PRIMARY OUTCOMES:
Percent change (%) from baseline in Non-HDL-C | at Week 8
  Percent change (%) from baseline at Week 8 in Non-HDL-C

SECONDARY OUTCOMES:
Percent change (%) from baseline in Non-HDL-C | Week 4
  Percent change (%) from baseline at Week 4 in Non-HDL-C
◦Percent change (%) from baseline at Week 4 and Week 8 in TG | Week 4 and Week 8
  Percent change (%) from baseline at Week 4 and Week 8 in TG
Percent change (%) from baseline at Week 4 and Week 8 in TC | Week 4 and Week 8
  Percent change (%) from baseline at Week 4 and Week 8 in TC
Percent change (%) from baseline at Week 4 and Week 8 in LDL-C | Week 4 and Week 8
  Percent change (%) from baseline at Week 4 and Week 8 in LDL-C
Percent change (%) from baseline at Week 4 and Week 8 in HDL-C | Week 4 and Week 8
  Percent change (%) from baseline at Week 4 and Week 8 in HDL-C
Percent change (%) from baseline at Week 4 and Week 8 in Apo A-I | Week 4 and Week 8
  Percent change (%) from baseline at Week 4 and Week 8 in Apo A-I
Percent change (%) from baseline at Week 4 and Week 8 in Apo B | Week 4 and Week
  Percent change (%) from baseline at Week 4 and Week 8 in Apo B

CONTACTS AND LOCATIONS:
Overall Officials: Hyo-Soo Kim, M.D., Principal Investigator — Seoul National University Hospital, Department of Internal Medicine
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No